CLINICAL TRIAL: NCT04229745
Title: Clinical Trial of Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) Oxygen in Women Having Planned Caesarean Delivery
Acronym: THRIVEN90
Status: Completed | Type: Observational
Sponsor: SABA AL-SULTTAN (Other)
Responsible Party: Sponsor-Investigator, SABA AL-SULTTAN, Research fellow, University College London Hospitals
Organization: University College London Hospitals (Other)
Other Study IDs: 18/0042
Record Dates: First submitted 2019-11-26; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Pre-oxygenation in Term Pregnant Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: THRIVE pre-oxygenation — Clinical Trial of Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) Oxygen in Women having Planned Caesarean Delivery

SUMMARY:
Clinical Trial of Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) Oxygen in Women having Planned Caesarean Delivery. Cohort study investigating the efficacy of THRIVE pre-oxygenation using pre-determined number of vital capacity breaths and comparing the efficacy to face mask pre-oxygenation. Aimed to recruit ASA 1-2 term pregnant women having elective caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo elective caesarean delivery
* singleton pregnancy
* American Society of Anaesthesiologists (ASA) Physical Status Grade II
* gestational age between 37 - 42 weeks

Exclusion Criteria:

* multiple pregnancy
* pre-eclampsia
* known fetal abnormality
* maternal cardio-respiratory comorbidity
* Body Mass Index (BMI) > 35 kg/m2.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: term pregnant women undergoing elective Caesarean section
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-06-23 (Actual); Study Completion 2019-06-23 (Actual)

PRIMARY OUTCOMES:
Number of vital capacity breaths required using THRIVE to pre-oxygenate 90% of parturients to an end tidal oxygen concentration of ≥90% (EN90). End tidal oxygen concentration >= 0.9 | 8 months study period
  measure end tidal oxygen concentration through breathing system attached to anaesthetic machine

SECONDARY OUTCOMES:
EN90 using THRIVE with mouth open versus mouth closed | 8 months study period
  to measure any difference in end tidal oxygen concentration after using THRIVE mouth closed versus THRIVE mouth open
comfort score of THRIVE | 8 months study period
  using 4-point Likert scale (1 being very uncomfortable- 4 comfortable)
changes in fetal wellbeing during pre-oxygenation time | 8 months study period
  using fetal cardiotocography

CONTACTS AND LOCATIONS:
Locations (1):
- UCLH, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided